CLINICAL TRIAL: NCT06046573
Title: Pilot Study of Internet-Delivered Psychological Treatment for Cancer Survivors With Clinically Significant Psychiatric Symptoms
Brief Title: Pilot Study of Internet-Delivered Psychological Treatment for Cancer Survivors
Acronym: IN-FACT-0
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Erland Axelsson, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-04056-01 #1
Record Dates: First submitted 2023-09-06; First posted 2023-09-21 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Cancer Survivors; Anxiety; Depression
Keywords: psycho-oncology; randomized factorial trial; Internet-delivered cognitive behavior therapy
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Internet-delivered psychological treatment, arm #1 (Experimental): Support and information + Behavioral activation
  Interventions: Behavioral: Support and information; Behavioral: Behavioral activation
- Internet-delivered psychological treatment, arm #2 (Experimental): Support and information + Systematic exposure with mindfulness training
  Interventions: Behavioral: Support and information; Behavioral: Systematic exposure with mindfulness training
- Internet-delivered psychological treatment, arm #3 (Experimental): Support and information + Promotion of health behaviors
  Interventions: Behavioral: Support and information; Behavioral: Promotion of health behaviors
- Internet-delivered psychological treatment, arm #4 (Experimental): Support and information + Behavioral activation + Systematic exposure with mindfulness training
  Interventions: Behavioral: Support and information; Behavioral: Behavioral activation; Behavioral: Systematic exposure with mindfulness training
- Internet-delivered psychological treatment, arm #5 (Experimental): Support and information + Behavioral activation + Promotion of health behaviors
  Interventions: Behavioral: Support and information; Behavioral: Behavioral activation; Behavioral: Promotion of health behaviors
- Internet-delivered psychological treatment, arm #6 (Experimental): Support and information + Systematic exposure with mindfulness training + Promotion of health behaviors
  Interventions: Behavioral: Support and information; Behavioral: Systematic exposure with mindfulness training; Behavioral: Promotion of health behaviors
- Internet-delivered psychological treatment, arm #7 (Experimental): Support and information + Behavioral activation + Systematic exposure with mindfulness training + Promotion of health behaviors
  Interventions: Behavioral: Support and information; Behavioral: Behavioral activation; Behavioral: Systematic exposure with mindfulness training; Behavioral: Promotion of health behaviors
- Internet-delivered psychological treatment, arm #8 (Experimental): Support and information
  Interventions: Behavioral: Support and information

INTERVENTIONS:
Behavioral: Support and information — Emotional and technical support. Information about the long-term effects of cancer.
Behavioral: Behavioral activation — Behavioral activation with existential themes and emphasis on values and relationships.
  Arms: Internet-delivered psychological treatment, arm #1; Internet-delivered psychological treatment, arm #4; Internet-delivered psychological treatment, arm #5; Internet-delivered psychological treatment, arm #7
Behavioral: Systematic exposure with mindfulness training — Systematic exposure with mindfulness training with a focus on anxiety about health and/or death, body image, and cancer-related trauma.
  Arms: Internet-delivered psychological treatment, arm #2; Internet-delivered psychological treatment, arm #4; Internet-delivered psychological treatment, arm #6; Internet-delivered psychological treatment, arm #7
Behavioral: Promotion of health behaviors — An overview of self-management techniques in terms of physical exercise, dietary advice, and strategies for improved sleep.
  Arms: Internet-delivered psychological treatment, arm #3; Internet-delivered psychological treatment, arm #5; Internet-delivered psychological treatment, arm #6; Internet-delivered psychological treatment, arm #7

SUMMARY:
Negative psychological effects of cancer are common, but cancer survivors are rarely offered structured psychological treatment. Internet-delivered treatments have shown some promise, but specific treatment components have not been empirically evaluated which means that it is not clear which therapies that should be prioritized. In this factorial pilot study, 48 cancer survivors with psychiatric symptoms are enrolled in variations on a 10-week therapist-guided online psychological treatment intended to address common negative psychological long-term effects of cancer. The aim of this study is to assess the feasibility of the study design and online treatment format. Key feasibility outcomes include interest in the study, patient-reported credibility of the intervention, adherence to the treatment protocol, satisfaction with the treatment, acceptability of the measurement strategy, missing data rates, adverse events, and preliminary efficacy on anxiety, depression, the fear of recurrence, and health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Cancer survivor at least 0.5 years after main therapy. Survivor of breast cancer (n=24), testicular cancer (n=12), or thyroid cancer (n=12).
* Clinically significant anxiety or depression (Patient Health Questionnaire 9 [PHQ-9]≥10, or Generalized Anxiety Disorder 7 [GAD-7]≥8, or 9-item Fear of Cancer Recurrence Inventory [FCRI-9]≥16)
* At least 18 years old
* Resident of Sweden (listed and de facto)
* Sufficient technical knowledge and knowledge of the Swedish language to take part in a text-based online treatment
* Continuous access to an electronic device that can be used to access the study web platform

Exclusion Criteria:

* Recurrent thoughts of suicide, as based on clinical judgement aided by the structured interview and the self-report version of the Montgomery-Åsberg Depression Rating Scale (MADRS-S) item 9
* Severe medical condition (e.g., very poor prognosis, stage IV cancer), severe psychiatric disorder (e.g., psychotic disorder, bipolar disorder, or severely debilitating substance use disorder, severe depression), or medical treatment (e.g., chemotherapy, immunotherapy, radiotherapy) that makes the treatment unfeasible
* Other ongoing psychological treatment
* Continuous psychotropic medication not stable for the past 4 weeks, or not expected to remain stable during the treatment period
* Planned absence for more than one week of the intended treatment period
* No complete the pre-treatment assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-03-10 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2024-10-22 (Actual)

PRIMARY OUTCOMES:
Feasibility 1: Feasibility of the randomized factorial design | Post-treatment assessment (immediately after treatment, completed within 45 days)
  A key feasibility outcome of this pilot study is the overall experience of study administrators and therapists tasked with the assignment and delivery of treatment variants in accordance with the randomized factorial design. After the main phase, all study administrators and therapists will be asked to rate the feasibility of the planned study design from 0 ("not feasible at all") to 10 ("fully feasible"), which will reported as a mean (SD) and median.
Feasibility 2: Credibility of the treatment as perceived by patients | Week 2 of treatment
  Credibility/Expectancy scale (C/E scale). Theoretical range: 0-50, where a higher score indicates higher credibility/expectancy.
Feasibility 3: Adherence to the treatment protocol #1 | Over the 10-week treatment period, with registration at the post-treatment assessment (immediately after treatment).
  Number of modules initiated, as registered by the clinician.
Feasibility 4: Adherence to the treatment protocol #2 | Each week from the beginning of treatment to the post-treatment assessment (immediately after treatment, completed within 45 days)
  Number of completed exercises, as based on a short weekly questionnaire tailored to suit each treatment arm, with corresponding questions about the number of days devoted to exposure exercises, days devoted to activity planning, and days devoted to the promotion of health behaviors.
Feasibility 5: Acceptability of the online measurement strategy #1 | Each week from the Each week from the beginning of treatment to the follow-up assessment (3 months after treatment)
  Number of measurements completed at each measurement point after the pre-treatment assessment. Preregistered target: at least 70% non-missing at the post-treatment and follow-up assessments.
Feasibility 6: Acceptability of the online measurement strategy #2 | Post-treatment assessment (within 45 days after treatment)
  Perceived strain caused by the measurement strategy. Preregistered target: at least 75% with a rating below 7 from 0 ("not at all stressful/distressing") to 10 ("extremely stressful/distressing").
Feasibility 7: Patients' satisfaction with the treatment #1 | Post-treatment assessment (within 45 days after treatment)
  The 8-item Client Satisfaction Questionnaire (CSQ-8). Theoretical range: 8-32, where a higher score indicates higher satisfaction.
Feasibility 8: Patients' satisfaction with the treatment #2 | Post-treatment assessment (within 45 days after treatment)
  Likert items pertaining to satisfaction with components.
Feasibility 9: Rate of adverse events and negative experiences #1 | Post-treatment assessment (within 45 days after treatment)
  Questionnaire used in previous clinical trials (e.g., ClinicalTrials.gov: NCT04511286)
Feasibility 10: Rate of adverse events and negative experiences #2 | Post-treatment assessment (within 45 days after treatment)
  20-item Negative Effects Questionnaire (NEQ-20). This will be reported as the proportion of endorsed items in the following subdomains: increase in symptoms, perceived insufficient quality of treatment, dependency, stigma, and hopelessness.
Feasibility 11: Preliminary efficacy in terms of within-group average change in general anxiety | Pre-treatment assessment (within 2 weeks before treatment) to post-treatment assessment (immediately after treatment, completed within 45 days)
  General Anxiety Disorder 7 (GAD-7, theoretical range: 0-21, where a higher score indicates more general anxiety)
Feasibility 12: Preliminary efficacy in terms of within-group average change in depressive symptoms | Pre-treatment assessment (within 2 weeks before treatment) to post-treatment assessment (immediately after treatment, completed within 45 days)
  Patient Health Questionnaire 9 (PHQ-9, theoretical range: 0-27, where a higher score indicates more symptoms of depression)
Feasibility 13: Preliminary efficacy in terms of within-group improvement in the fear of cancer recurrence | Pre-treatment assessment (within 2 weeks before treatment) to post-treatment assessment (immediately after treatment, completed within 45 days)
  9-item Fear of Cancer Recurrence Inventory (FCRI-9, theoretical range: 0-36, where a higher score indicates a more pronounced fear of cancer recurrence)
Feasibility 14: Preliminary efficacy in terms of within-group improvement in health-related quality of life | Pre-treatment assessment (within 2 weeks before treatment) to post-treatment assessment (immediately after treatment, completed within 45 days)
  36-item Short Form Health Survey (SF-36, scored as a Mental Health Component Score and a Physical Health Component Score according to standard norms, both with a theoretical range of 0-100, where a higher score indicates a higher health-related quality of life)

SECONDARY OUTCOMES:
Symptom domains surveyed primarily to assess the feasibility of the measurement method: Health anxiety. | Pre-treatment assessment (within 2 weeks before treatment) to post-treatment assessment (immediately after treatment, completed within 45 days). Secondary analysis: from pre-treatment up to follow-up 3 months after treatment.
  14-item Health Anxiety Inventory (HAI-14, theoretical range: 0-42, where a higher score indicates more health anxiety).
Symptom domains surveyed primarily to assess the feasibility of the measurement method: Somatic symptom burden. | Pre-treatment assessment (within 2 weeks before treatment) to post-treatment assessment (immediately after treatment, completed within 45 days). Secondary analysis: from pre-treatment up to follow-up 3 months after treatment.
  Somatic Symptom Scale 8 (SSS-8, theoretical range: 0-32, where a higher score indicates a higher somatic symptom burden). Exploratory secondary analyses will be based on individual items, each scored 0-4.
Symptom domains surveyed primarily to assess the feasibility of the measurement method: Body image distress. | Screening (within 6 months before treatment) to post-treatment assessment (immediately after treatment, completed within 45 days).
  Body Image Scale (BIS, theoretical range: 0-30, where a higher score indicates a higher level of body image distress).
Symptom domains surveyed primarily to assess the feasibility of the measurement method: Disability. | Pre-treatment assessment (within 2 weeks before treatment) to post-treatment assessment (immediately after treatment, completed within 45 days). Secondary analysis: from pre-treatment up to follow-up 3 months after treatment.
  12-item WHO Disability Assessment Schedule 2.0 (WD2-12, theoretical range: 0-100, where a higher score indicates more disability).
Process and target variables surveyed primarily to assess the feasibility of the measurement method: Behavioral activation | Pre-treatment (within 2 weeks before treatment), once each week during treatment (9 assessments in total), post-treatment (after treatment, completed within 45 days), and at follow-up 3 months after treatment (completed within 45 days).
  3-item Behavioral Activation for Depression Scale - Activation (BADS-AC-3, theoretical range: 0-18, where a higher score indicates a higher level of behavioral activation).
Process and target variables surveyed primarily to assess the feasibility of the measurement method: Symptom preoccupation | Pre-treatment (within 2 weeks before treatment), once each week during treatment (9 assessments in total), post-treatment (after treatment, completed within 45 days), and at follow-up 3 months after treatment (completed within 45 days).
  Symptom Preoccupation Scale (preliminary scale). A higher score indicates higher degree of preoccupation with symptoms. This is to be regarded as an an item pool, and the scale is is under development, which means that the total range cannot be preregistered.
Process and target variables surveyed primarily to assess the feasibility of the measurement method: Physical activity | Pre-treatment (within 2 weeks before treatment), once each week during treatment (9 assessments in total), post-treatment (after treatment, completed within 45 days), and at follow-up 3 months after treatment (completed within 45 days).
  Godin-Shephard Leisure-Time Physical Activity Questionnaire (GSLTPAQ, theoretical range 0-99, where a higher score indicates a higher level of physical activity). If necessary for statistical modeling, the GSLTPAQ will be dichotomized to indicate active (≥24) vs. insufficiently active (<24).
Process and target variables surveyed primarily to assess the feasibility of the measurement method: Health-related self-efficacy. | Pre-treatment (within 2 weeks before treatment), once each week during treatment (9 assessments in total), post-treatment (after treatment, completed within 45 days), and at follow-up 3 months after treatment (completed within 45 days).
  Based loosely on the Arthritis Self-efficacy Scale. Theoretical range of 0-60, where a higher score indicates a higher level of general health-related self-efficacy.
Relationship with the therapist (therapeutic alliance) | Week 2 of treatment
  Working Alliance Inventory (WAI, theoretical range: 6-42, where a higher score indicates a stronger therapeutic alliance)
Screening only: Alcohol use | At screening
  Alcohol Use Disorders Identification Test (AUDIT, theoretical range: 0-40, where a higher score indicates more problematic alcohol use).
Screening only: Substance use | At screening
  Drug Use Disorders Identification Test (DUDIT, theoretical range: 0-44, where a higher score indicates more problematic substance use).
Screening only: General distress | At screening
  Hospital Anxiety and Depression Scale (HADS, theoretical range: 0-42, where a higher score indicates more general distress).

CONTACTS AND LOCATIONS:
Overall Officials: Erland Axelsson, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Individual participant data from this pilot study fall under Swedish and European Union data protection and privacy legislation and can therefore not be share in their entirety. Reasonable requests may be directed to the corresponding author, and will be considered on a case-by-case basis.

REFERENCES:
- [Derived] Winter J, Gasslander N, Rane G, Sundstrom F, Bjorkhem-Bergman L, Hedman C, Axelsson E. Proof-of-concept for a randomized factorial design strategy to build a complex online support program for cancer survivors with psychiatric symptoms: the IN-FACT-0 feasibility trial. J Cancer Surviv. 2025 Oct 25. doi: 10.1007/s11764-025-01905-2. Online ahead of print. PMID 41136825

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-16): https://cdn.clinicaltrials.gov/large-docs/73/NCT06046573/Prot_SAP_000.pdf